CLINICAL TRIAL: NCT00493623
Title: A Randomized, Double-blind Study of the Efficacy of Intravenous Bonviva in the Relief of Pain After Recent Vertebral Osteoporotic Fracture in Osteoporotic Patients.
Brief Title: BONDIR Study: A Study of Intravenous Bonviva (Ibandronate) After Recent Vertebral Osteoporotic Fracture in Patients With Osteoporosis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ML19360
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-03

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Ibandronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: ibandronate [Bonviva/Boniva]
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo i.v. single dose
  Arms: 2
Drug: ibandronate [Bonviva/Boniva] — 3mg i.v. single dose
  Arms: 1

SUMMARY:
This 2 arm study will assess the efficacy and safety of intravenous Bonviva in patients with osteoporosis experiencing pain after recent vertebral osteoporotic fracture. Patients will be randomized to receive either Bonviva (3mg i.v. bolus injection) or placebo. The anticipated time on study treatment is <3 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women or men >30 years of age;
* osteoporosis;
* vertebral osteoporotic fracture in past 4 weeks;
* fracture-related pain requiring analgesic treatment.

Exclusion Criteria:

* non-menopausal women;
* current treatment with another bisphosphonate;
* current treatment with class III analgesics.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2007-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Success of Bonviva therapy (>=20% diminution of pain intensity between day 0 and 7, with stabilization or diminution of concomitant analgesics between day 3 and 7). | Day 7

SECONDARY OUTCOMES:
Percentage of patients with >=50% diminution of pain between day 0 and 7 | Day 7
Pain control | Day 7 and 1 month
Analgesic medication | 1 month
Hospitalization | 1 month
AEs and laboratory parameters | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (22):
- France (22):
  - Aix-en-Provence
  - Amiens
  - Angers
  - Bonneville
  - Bordeaux
  - Caen
  - Cannes
  - Clermont-Ferrand
  - Échirolles
  - Lille
  - Lomme
  - Marseille
  - Montpellier
  - Mulhouse
  - Nantes
  - Nice
  - Orléans
  - Paris
  - Rennes
  - Rouen
  - Saint-Priest-en-Jarez
  - Toulouse